CLINICAL TRIAL: NCT01358175
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Secukinumab to Demonstrate the 16 Week Efficacy and to Assess the Long Term Safety, Tolerability and Efficacy up to 2 Years in Patients With Active Ankylosing Spondylitis
Brief Title: 16 Week Efficacy and 2 Year Long Term Safety and Efficacy of Secukinumab in Patients With Active Ankylosing Spondylitis
Acronym: MEASURE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2305; 2010-024529-18 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; AS; ASAS; inflammatory back pain
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Secukinumab 10 mg/kg i.v. / 75 mg s.c. (Experimental): Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection every four weeks until the end of the study.
  Interventions: Drug: Secukinumab (75 mg)
- Secukinumab 10 mg/kg i.v. / 150 mg s.c. (Experimental): Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection every four weeks until the end of the study.
  Interventions: Drug: Secukinumab (150 mg)
- Placebo (Placebo Comparator): Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection every four weeks until the end of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab (75 mg) — Secukinumab (75 mg)
  Arms: Secukinumab 10 mg/kg i.v. / 75 mg s.c.
Drug: Secukinumab (150 mg) — Secukinumab (150 mg)
  Arms: Secukinumab 10 mg/kg i.v. / 150 mg s.c.
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of secukinumab in patients with active ankylosing spondylitis who are intolerant to or have had an inadequate response to NSAIDs, DMARDs and / or TNFα inhibitor therapy.

ELIGIBILITY:
Inclusion criteria:

* Male or non-pregnant, non-lactating female patients at least 18 years of age
* Diagnosis of moderate to severe AS with prior documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984)
* Patients should have been on NSAIDs with an inadequate response
* Patients who are regularly taking NSAIDs as part of their AS therapy are required to be on a stable dose
* Patients who have been on an anti-TNFα agent (not more than one) must have experienced an inadequate response

Exclusion criteria:

* Chest X-ray with evidence of ongoing infectious or malignant process
* Patients with total ankylosis of the spine
* Patients previously treated with any biological immunomodulating agents except for those targeting TNFα
* Previous treatment with any cell-depleting therapies
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (63):
- United States (10):
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Cedar Rapids, Iowa
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Benbrook, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Spokane, Washington
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Bulgaria (3):
  - Novartis Investigative Site, Burgas, Bulgaria
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
- Canada (3):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Toronto, Ontario
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Paris
- Germany (9):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ratingen
- Italy (6):
  - Novartis Investigative Site, Valeggio sul Mincio, (vr)
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
- Mexico (4):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacán, Sinaloa
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Peru (5):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, La Victoria, Lima region
  - Novartis Investigative Site, Pueblo Libre, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Surquillo, Lima region
- Russia (5):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Taiwan (2):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Gaziantep
- United Kingdom (4):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Jamaludin A, Windsor R, Ather S, Kadir T, Zisserman A, Braun J, Gensler LS, Ostergaard M, Poddubnyy D, Coroller T, Porter B, Ligozio G, Readie A, Machado PM. Automated detection of spinal bone marrow oedema in axial spondyloarthritis: training and validation using two large phase 3 trial datasets. Rheumatology (Oxford). 2025 Oct 1;64(10):5446-5454. doi: 10.1093/rheumatology/keaf323. PMID 40489668
- [Derived] Braun J, Buehring B, Baraliakos X, Gensler LS, Porter B, Quebe-Fehling E, Haemmerle S. Effects of secukinumab on bone mineral density and bone turnover biomarkers in patients with ankylosing spondylitis: 2-year data from a phase 3 study, MEASURE 1. BMC Musculoskelet Disord. 2021 Dec 13;22(1):1037. doi: 10.1186/s12891-021-04930-1. PMID 34903218
- [Derived] van der Horst-Bruinsma I, Miceli-Richard C, Braun J, Marzo-Ortega H, Pavelka K, Kivitz AJ, Deodhar A, Bao W, Porter B, Pournara E. A Pooled Analysis Reporting the Efficacy and Safety of Secukinumab in Male and Female Patients with Ankylosing Spondylitis. Rheumatol Ther. 2021 Dec;8(4):1775-1787. doi: 10.1007/s40744-021-00380-2. Epub 2021 Oct 7. PMID 34618347
- [Derived] Schett G, Baraliakos X, Van den Bosch F, Deodhar A, Ostergaard M, Gupta AD, Mpofu S, Fox T, Winseck A, Porter B, Shete A, Gensler LS. Secukinumab Efficacy on Enthesitis in Patients With Ankylosing Spondylitis: Pooled Analysis of Four Pivotal Phase III Studies. J Rheumatol. 2021 Aug;48(8):1251-1258. doi: 10.3899/jrheum.201111. Epub 2021 Mar 15. PMID 33722947
- [Derived] Baraliakos X, Van den Bosch F, Machado PM, Gensler LS, Marzo-Ortega H, Sherif B, Quebe-Fehling E, Porter B, Gaillez C, Deodhar A. Achievement of Remission Endpoints with Secukinumab Over 3 Years in Active Ankylosing Spondylitis: Pooled Analysis of Two Phase 3 Studies. Rheumatol Ther. 2021 Mar;8(1):273-288. doi: 10.1007/s40744-020-00269-6. Epub 2020 Dec 22. PMID 33351179
- [Derived] Himmler S, Branner JC, Ostwald DA. The societal impact of a biologic treatment of ankylosing spondylitis: a case study based on secukinumab. J Comp Eff Res. 2021 Feb;10(2):143-155. doi: 10.2217/cer-2020-0077. Epub 2020 Nov 30. PMID 33252266
- [Derived] Kvien TK, Conaghan PG, Gossec L, Strand V, Ostergaard M, Poddubnyy D, Williams N, Porter B, Shete A, Gilloteau I, Deodhar A. Secukinumab and Sustained Reduction in Fatigue in Patients With Ankylosing Spondylitis: Long-Term Results of Two Phase III Randomized Controlled Trials. Arthritis Care Res (Hoboken). 2022 May;74(5):759-767. doi: 10.1002/acr.24517. Epub 2022 Mar 10. PMID 33227175
- [Derived] Deodhar AA, Miceli-Richard C, Baraliakos X, Marzo-Ortega H, Gladman DD, Blanco R, Das Gupta A, Martin R, Safi J Jr, Porter B, Shete A, Rosenbaum JT. Incidence of Uveitis in Secukinumab-treated Patients With Ankylosing Spondylitis: Pooled Data Analysis From Three Phase 3 Studies. ACR Open Rheumatol. 2020 May;2(5):294-299. doi: 10.1002/acr2.11139. Epub 2020 Apr 30. PMID 32352653
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Braun J, Deodhar A, Landewe R, Baraliakos X, Miceli-Richard C, Sieper J, Quebe-Fehling E, Martin R, Porter B, Gandhi KK, van der Heijde D; MEASURE 1 and MEASURE 2 study groups. Impact of baseline C-reactive protein levels on the response to secukinumab in ankylosing spondylitis: 3-year pooled data from two phase III studies. RMD Open. 2018 Nov 21;4(2):e000749. doi: 10.1136/rmdopen-2018-000749. eCollection 2018. PMID 30564451
- [Derived] Wei JC, Baeten D, Sieper J, Deodhar A, Bhosekar V, Martin R, Porter B. Efficacy and safety of secukinumab in Asian patients with active ankylosing spondylitis: 52-week pooled results from two phase 3 studies. Int J Rheum Dis. 2017 May;20(5):589-596. doi: 10.1111/1756-185X.13094. Epub 2017 May 25. PMID 28544533
- [Derived] Braun J, Baraliakos X, Deodhar A, Baeten D, Sieper J, Emery P, Readie A, Martin R, Mpofu S, Richards HB; MEASURE 1 study group. Effect of secukinumab on clinical and radiographic outcomes in ankylosing spondylitis: 2-year results from the randomised phase III MEASURE 1 study. Ann Rheum Dis. 2017 Jun;76(6):1070-1077. doi: 10.1136/annrheumdis-2016-209730. Epub 2016 Dec 13. PMID 27965257
- [Derived] Deodhar AA, Dougados M, Baeten DL, Cheng-Chung Wei J, Geusens P, Readie A, Richards HB, Martin R, Porter B. Effect of Secukinumab on Patient-Reported Outcomes in Patients With Active Ankylosing Spondylitis: A Phase III Randomized Trial (MEASURE 1). Arthritis Rheumatol. 2016 Dec;68(12):2901-2910. doi: 10.1002/art.39805. PMID 27390130
- [Derived] Baeten D, Sieper J, Braun J, Baraliakos X, Dougados M, Emery P, Deodhar A, Porter B, Martin R, Andersson M, Mpofu S, Richards HB; MEASURE 1 Study Group; MEASURE 2 Study Group. Secukinumab, an Interleukin-17A Inhibitor, in Ankylosing Spondylitis. N Engl J Med. 2015 Dec 24;373(26):2534-48. doi: 10.1056/NEJMoa1505066. PMID 26699169

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo iv at baseline, Week 2 and Week 4, and then placebo sc at Week 8 and Week 12
Period: Overall Study
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Started | 124 | 125 | 122
Completed | 103 | 97 | 90
Not Completed | 21 | 28 | 32
Not completed — Death | 1 | 0 | 1
Not completed — Withdrawal by Subject | 9 | 5 | 10
Not completed — Technical issues | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Non Compliance with Study Treatment | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Lack of Efficacy | 3 | 8 | 6
Not completed — Adverse Event | 6 | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo | Total
Number analyzed (Participants) | 124 | 125 | 122 | 371
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 117 | 122 | 115 | 354
  >=65 years | 7 | 3 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 37 | 114
  Male | 88 | 84 | 85 | 257

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Responders for the SpondyloArthritis International Society / ASAS 20 Response
Description: ASAS 20 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined timeframe at least 20% improvement in score in at least 3 of a conventional set of 4 clinical domains relevent to AS and no worsening in the fourth domain. ASAS 20 is used to assess the efficacy of at least one dose of secukinumab against placebo.
Time Frame: 16 weeks
Population: FAS comprised all patients who were randomized and to whom study treatment had been assigned. The efficacy analyses are based on the FAS.
Measure: Number; unit: % responders
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
% responders | 59.7 | 60.8 | 28.7
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 75 mg s.c. vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.76, 95% CI 2-sided [2.20 to 6.42]
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.89, 95% CI 2-sided [2.28 to 6.65]

2. Secondary Outcome: Assessment of Responders for the SpondyloArthritis International Society ASAS 40 Response
Description: ASAS 40 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined timeframe at least 40% improvement in score in at least 3 of a conventional set of 4 clinical domains relevent to AS and no worsening in the fourth domain. ASAS 40 is used to assess the efficacy of at least one dose of secukinumab against placebo.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Number; unit: % responders
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
% responders | 33.1 | 41.6 | 13.1

3. Secondary Outcome: Change From Baseline in Serum hsCRP
Description: The change from baseline in hsCRP is expressed as a ratio of post-baseline to baseline values. With the ratio normalized to 1.0 at baseline, ratios less than 1.0 represent decreased postbaseline values, whereas ratios greater than 1.0 represent increased post-baseline values.
Time Frame: Base line and Week 16
Population: FAS. Analysis was done on the log(e) ratio of the treatment value vs. baseline value to normalize the distribution of the hsCRP at each visit. LS Mean, SE, 95% CI and p-value are from mixed-effect model repeated measures (MMRM) with treatment, visit, TNF-alpha inhibitor status as factors, log(e) baseline and weight as covariates.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
ratio | 0.45 (1.092) | 0.4 (1.090) | 0.97 (1.095)

4. Secondary Outcome: Assessment of Responders for the SpondyloArthritis International Society ASAS 5/6 Response
Description: ASAS 5/6 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined timeframe at least 20% improvement in score in at least 5 of a conventional set of 6 clinical domains relevent to AS and no worsening in the remaining domain. In this study, ASAS 5/6 is used to assess the efficacy of at least one dose of secukinumab against placebo.
Time Frame: 16 weeks
Measure: Number; unit: % responders
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
% responders | 45.2 | 48.8 | 13.1

5. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index / BASDAI
Description: BASDAI is a validated assessment tool using 0 through 10 scales (0 indicating "no problem" and 10 indicating " worst problem"), to characterize six clinical domains pertaining to five major symptoms of AS perceived by the patients. Computed composite scores of 4 or greater indicate suboptimal disease control. In this study, the BASDAI is used to assess the efficacy of at least one dose of secukinumab verus placebo. To give each symptom equal weighting, the mean (average) of the two scores relating to morning stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score. Scores of 4 or greater suggest suboptimal control of disease, and patients with scores of 4 or greater are usually good candidates for either a change in their medical therapy or for enrollment in clinical trials evaluating new drug therapies directed at Ankylosing Spondylitis.
Time Frame: Baseline and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
units on scale | -2.34 (0.175) | -2.32 (0.172) | -0.59 (0.180)

6. Secondary Outcome: Change From Baseline in Physical Function Component of the Short-form Health Survey / SF-36 PCS
Description: SF-36 is a 36 item questionnaire which measures Quality of Life across eight domains, which are both phyically and emotionally based. Two overall summary scores, the Phyical Component Summary (PCS) and Mental Component Summary (MCS) can be computed. In this study, SF-36 PCS is used to assess improvement from baseline of at least one dose of secukinumab versus placebo.The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: baseline, 16 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
units on a scale | 5.64 (0.595) | 5.57 (0.586) | 0.96 (0.612)

7. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life Questionnaire / ASQoL
Description: ASQoL is an 18 item questionnaire that assesses disease-specific quality of life (QoL), consisting of statements that are relevant to the physical and mental conditions for a participant with AS: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each statement is answered by the participant as a 'Yes' (scored as 1) or 'No' (scored as 0). All item scores are summed to give a total score. Total score can range from 0 (good QoL) to 18 (poor QoL). In this study, ASQoL is used to assess improvement from baseline of at least one dose of secukinumab versus placebo.
Time Frame: baseline and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
units on a scale | -3.61 (0.424) | -3.58 (0.420) | -1.04 (0.437)

8. Secondary Outcome: Assessment of Responders for ASAS Partial Remission
Description: ASAS partial remission is a composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame a value not above 2 units in each of the 4 ASAS domains on a scale of 10. In this study ASAS partial remission is used to assess the efficacy of at least one dose of secukinumab versus placebo.ASAS partial remission was defined as a VAS score of less than 2 units in each of the 4 domains of ASAS 20: participant global assessment, pain (total back pain), function and inflammation. The percentages of participants who achieved ASAS partial remission were calculated.
Time Frame: 16 weeks
Measure: Number; unit: % responders
Arm/Group | Secukinumab 10 mg/kg i.v. / 75 mg s.c. | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Placebo
Number analyzed (Participants) | 124 | 125 | 122
% responders | 16.1 | 15.2 | 3.3

ADVERSE EVENTS:
Time Frame: Baseline to week 104
Description: Patients initially randomized to placebo were assessed for ASAS 20 response at Week 16 and switched to active treatment at Week 16 (for placebo non-responders) or at Week 24 (for placebo responders). Blinding was maintained beyond the primary endpoint to ensure reliable efficacy and safety measures
Groups:
- Secukinumab 10mg/kg -75 mg; Secukinumab 10mg/kg -150 mg: Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection every four weeks until the end of the study.
- Placebo Secukinumab: Placebo iv at baseline, Week 2 and Week 4, and then placebo sc at Week 8 and Week 12 up to end of Study
- Placebo Non-Resp Secukinumab 75 mg: Placebo iv at baseline, Week 2 and Week 4, and then placebo sc at Week 8 and Week 12 re-randomized non-responder week 16 to Secukinumab 75 mg
- Placebo Non-Resp Secukinumab 150 mg: Placebo iv at baseline, Week 2 and Week 4, and then placebo sc at Week 8 and Week 12 re-randomized non-responder week 16 to Secukinumab 150 mg
- Placebo Resp Secukinumab 75 mg: Placebo iv at baseline, Week 2 and Week 4, and then placebo sc at Week 8 and Week 12 re-randomized non-responder week 24 to Secukinumab 75 mg
- Placebo Resp Secukinumab 150 mg: Placebo iv at baseline, Week 2 and Week 4, and then placebo sc at Week 8 and Week 12 re-randomized non-responder week 24 to Secukinumab 150 mg
Arm/Group | Secukinumab 10mg/kg -75 mg | Secukinumab 10mg/kg -150 mg | Placebo Secukinumab | Placebo Non-Resp Secukinumab 75 mg | Placebo Non-Resp Secukinumab 150 mg | Placebo Resp Secukinumab 75 mg | Placebo Resp Secukinumab 150 mg
Serious Adverse Events (participants affected / at risk) | 16/124 | 13/125 | 5/122 | 5/39 | 8/38 | 3/17 | 1/18
Other Adverse Events (participants affected / at risk) | 88/124 | 100/125 | 52/122 | 24/39 | 27/38 | 12/17 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 10mg/kg -75 mg (N=124) | Secukinumab 10mg/kg -150 mg (N=125) | Placebo Secukinumab (N=122) | Placebo Non-Resp Secukinumab 75 mg (N=39) | Placebo Non-Resp Secukinumab 150 mg (N=38) | Placebo Resp Secukinumab 75 mg (N=17) | Placebo Resp Secukinumab 150 mg (N=18)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Application site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 10mg/kg -75 mg (N=124) | Secukinumab 10mg/kg -150 mg (N=125) | Placebo Secukinumab (N=122) | Placebo Non-Resp Secukinumab 75 mg (N=39) | Placebo Non-Resp Secukinumab 150 mg (N=38) | Placebo Resp Secukinumab 75 mg (N=17) | Placebo Resp Secukinumab 150 mg (N=18)
Leukopenia (Blood and lymphatic system disorders) | 10 | 8 | 1 | 1 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 3 | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0
Iritis (Eye disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0
Uveitis (Eye disorders) | 4 | 4 | 2 | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 8 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 9 | 7 | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 16 | 21 | 7 | 4 | 3 | 2 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 8 | 5 | 3 | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 8 | 2 | 2 | 1 | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 3 | 2 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 2 | 0 | 4 | 0 | 0
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 3 | 2 | 0 | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 6 | 2 | 0 | 2 | 1 | 2
Infection parasitic (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 7 | 12 | 2 | 4 | 4 | 2 | 1
Nasopharyngitis (Infections and infestations) | 25 | 34 | 9 | 7 | 6 | 3 | 4
Oral herpes (Infections and infestations) | 2 | 6 | 0 | 0 | 2 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 10 | 18 | 1 | 2 | 1 | 0 | 2
Rhinitis (Infections and infestations) | 4 | 8 | 0 | 1 | 3 | 0 | 1
Sinusitis (Infections and infestations) | 4 | 5 | 3 | 0 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 17 | 9 | 2 | 2 | 6 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 7 | 0 | 1 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 0 | 1 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 3 | 5 | 0 | 1 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 1 | 1 | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 1 | 0 | 1 | 0 | 1
Low density lipoprotein increased (Investigations) | 1 | 3 | 1 | 0 | 2 | 0 | 0
Osteoprotegerin decreased (Investigations) | 2 | 4 | 2 | 0 | 2 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 15 | 13 | 6 | 1 | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 11 | 4 | 3 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 11 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 2 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 2 | 1 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 1 | 1 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 6 | 4 | 1 | 1 | 0 | 1
Headache (Nervous system disorders) | 18 | 18 | 7 | 2 | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 2 | 5 | 0 | 1 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 2 | 1 | 1 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 2 | 2 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 6 | 3 | 4 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6 | 1 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 1 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 6 | 4 | 0 | 1 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.